CLINICAL TRIAL: NCT00440180
Title: The Role of Aromatase Inhibitors in the Treatment of Infertility in Obese Male
Brief Title: Aromatase Inhibitors in the Treatment of Male Infertility
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not able meet target enrollment.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00016246
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Obesity; Oligospermia
Keywords: Obesity; Low sperm count; Male infertility
MeSH Terms: conditions — Obesity; Oligospermia; Infertility, Male | interventions — Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Group A (Experimental): Anastrozole
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — 1 mg qd for 4 months
  Other Names: Arimidex
  Arms: Group A
Drug: Placebo — Placebo Comparator
  Arms: Group B

SUMMARY:
Obesity is associated with an increase in blood levels of estrogen. Estrogen or "female hormone" is believed to have a negative effect on sperm production. Aromatase inhibitors such as anastrozole work to decrease the production of estrogen and increase testosterone in the body. By decreasing the level of estrogen, sperm production should improve. In this study, the investigators will try to determine the benefit of anastrozole in obese men and follow pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male partner of a couple presenting for infertility work up after one year of unprotected intercourse
2. Moderate oligozoospermia (defined as mean sperm count ≤ 20 × 106/mL and ≥ than 3 × 106/mL) of at least two separate occasions spanning a minimum of two weeks
3. Obese men BMI ≥ 30
4. FSH and LH levels < 10 mIU/mL

Exclusion Criteria:

1. Severe Oligozoospermia: Sperm count < than 3 × 106/mL, including azoospermia
2. Age less than 18 or greater than 65 years
3. Pyospermia or leukospermia: defined by white blood cells ≥ 1 million leukocytes per milliliter of semen
4. Cryptorchidism
5. Vasectomy reversal
6. Regular use of tobacco products
7. BMI < 30
8. Use of anabolic steroids or testosterone replacement
9. All patients with abnormal initial liver function tests "AST or ALT" will be excluded form the study

Ages: 16 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad O Hammoud, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo once daily
- Anastrozole: 1 milligram daily
Period: Overall Study
Arm/Group | Placebo | Anastrozole
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Anastrozole | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate
Description: Partner pregnancy rate during study participation
Time Frame: 4 months
Measure: Number; unit: participants partner
Arm/Group | Placebo | Anastrozole
Number analyzed (Participants) | 10 | 10
participants partner | 0 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Anastrozole
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 3/20 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Anastrozole (N=10)
Axillary Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Anastrozole (N=20)
Increased Liver Enzymes (General disorders) | 2 (2) | 2 (2)
Headache (General disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No